CLINICAL TRIAL: NCT00555633
Title: Regular Use of an SPF30 Sunscreen and an After-sun-lotion in Skin Cancer Risk Patients, Particularly in Xeroderma Pigmentosum and Basal Cell Nevus Syndrome
Brief Title: Use of an SPF30 Sunscreen and an After-sun-lotion in Skin Cancer Risk Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Peter Wolf, MD, Principal Investigator, Medical University of Graz, Austria
Other Study IDs: 16-015 ex 04/05
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Skin Cancer; Xeroderma Pigmentosum; Basal Cell Nevus Syndrome
Keywords: Photoprotection; Sunscreen; After-sun-lotion; DNA repair enzymes; liposomes; skin cancer; Xeroderma pigmentosum; Basal cell nevus syndrome
MeSH Terms: conditions — Skin Neoplasms; Xeroderma Pigmentosum; Basal Cell Nevus Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Study aim: To determine the effect of an intensified daily photoprotection over 24 months with an SPF30 sunscreen and an after sun-lotion both containing liposomal DNA repair enzymes in a population of patients at high-risk for skin cancer, including xeroderma pigmentosum (XP) and basal cell nevus syndrome.

DETAILED DESCRIPTION:
An SPF 30 sunscreen and a proprietary after sun lotion both containing a combination of plankton extract and micrococcus lysate (kindly provided by ATEIA AG, Vaduz, Liechtenstein) was used in a pilot study of intensified photoprotection in patients with multiple skin cancers. Thirteen patients (8 women and 5 men), between 37 and 81 years old, who had had a history of multiple skin cancers were enrolled in the study. Five of the patients had xeroderma pigmentosum (XP) (complementation group: A, 2; C,1; and non-classified 2); one patient XP variant, 3 patients basal cell nevus syndrome, and four patients no skin cancer syndrome. Patients were instructed to apply their sunscreen regularly before sun exposure and 4.5 ml of the after sun lotion to their face and arms daily, as close to mid-day as possible for a period of up to 24 months. The patients were examined in 3-month intervals and the new appearance of actinic keratoses and skin cancers was recorded. New lesions were removed at these visits and the pathology was confirmed by histological examination, except in the cases of (multiple) actinic keratoses, whenever patients agreed. The number of skin tumors during the 24 months of the study was compared to the number in the preceding 24 month-period before study entry. The data were obtained from patient charts and/or electronic files. There was a statistical trend for less BCCs during the study period compared to the prestudy period. In addition, the patients received at each of the 3-month visits a questionnaire and were asked to rate the status of their skin on face and arms during the last 3 months for various parameters on a scale from -2 (maximum worsening) to +2 (maximum improvement). The patients' ratings revealed a statistically significant improvement for several parameters: smoothness, color spots, wrinkles, burning, irritation, teleangiectasia, infections, warts, and skin lesions or sores, starting as early than at the first 3-month visit with a maximum effect seen at 12 months. No adverse effects were noted during the study.

ELIGIBILITY:
Inclusion Criteria:

* Xeroderma pigmentosum
* Basal cell nevus syndrome
* Other patient with a history of multiple skin cancers (three or more lesions, including actinic keratosis, squamous cell carcinoma, basal cell carcinoma, and/or malignant melanoma)

Exclusion Criteria:

* Intolerance of study preparation
* Allergy against study preparation
* Non-acceptable side effects

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2004-10; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Number of skin cancers | retrospective

SECONDARY OUTCOMES:
Patients' skin score parameters (including smoothness, color spots, wrinkles, burning, irritation, teleangiectasia, infections, warts, and skin lesions or sores) | retrospective

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wolf, MD, Principal Investigator — Medical University of Graz, Austria
Locations (1):
- Medical University of Graz, Department of Dermatology, Graz, Austria